CLINICAL TRIAL: NCT05095636
Title: A Phase II Randomized Controlled Trial of Apatinib Monotherapy Versus Apatinib Combined With Camrelizumab in Third-line or Later-line Treatment of Advanced Gastric Adenocarcinoma
Brief Title: Apatinib Monotherapy Versus Apatinib Combined With Camrelizumab for Third-line Treatment of Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-CAP
Record Dates: First submitted 2021-10-02; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Gastric Cancer; Metastasis
Keywords: gastric cancer; target therapy; metastasis; apatinib; anti-PD-1 antibody
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apatinib monotherapy (Active Comparator): Apatinib，500 mg，po., qd, q2w
  Interventions: Drug: Apatinib Mesylate
- Apatinib Combined With Camrelizumab (Experimental): Apatnib，250 mg，po., qd，q2w; Camrelizumab，200mg， ivgtt，d1, q2w
  Interventions: Drug: Apatinib Mesylate; Drug: Camrelizumab

INTERVENTIONS:
Drug: Apatinib Mesylate — oral Apatinib once everyday
Drug: Camrelizumab — intravenous camrelizumab 200mg once every two weeks
  Arms: Apatinib Combined With Camrelizumab

SUMMARY:
This open, single-center, randomized phase II study was to evaluate the clinical benefit of apatinib plus camrelizumab which is an anti-Programmed cell death-1 (PD-1) monoclonal antibody, versus apatinib in patients with metastatic gastric cancer refractory to two or more lines of treatment, fully evaluating the efficacy and safety of the combined regimen.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignant tumors with the highest mortality in the world. Post-line treatment options for metastatic gastric cancer (mGC) are limited. Monoclonal antibodies targeting Vascular Endothelial Growth Factor Receptor 2 (VEGFR-2) and small molecule tyrosine kinase inhibitors (TKIs) have shown benefits on progression free survival (PFS) and overall survival (OS) in second-line or third-line treatment of mGC. Following a phase III randomized clinical trial, apatinib, an oral small-molecule drug targeted with VEGFR-2, has been proved to significantly prolong patients' OS in the third-line or later-line treatment of mGC, thus becoming the standard third-line or later-line regimen for gastric cancer in China. In immunotherapy of mGC, pembrolizumab has been approved for third-line treatment of programmed cell death-Ligand 1 (PD-L1) positive advanced gastric cancer, and nivolumab also become the standard third-line treatment regimen. What is the best option for third-line treatment of metastatic gastric cancer remains unclear. Analysis from the subgroup of the Attraction 2 study showed that patients who had previously been treated with anti-VEGFR targeted drug ramucizumab had significantly higher PFS and OS than those who had not. The REGONIVO study also showed that the anti-angiogenic TKI regorafenib combined with nivolumab achieved a good objective response rate after the failure of standard treatment in gastric cancer. Therefore, it is worth exploring whether apatinib combined with anti-PD-1 monoclonal antibody could bring improvements in PFS and OS while compared with apatinib monotherapy. This open, single-center, randomized phase II study was to evaluate the clinical benefit of apatinib plus camrelizumab which is an anti-PD-1 monoclonal antibody, versus apatinib in patients with metastatic gastric cancer refractory to two or more lines of treatment, fully evaluating the efficacy and safety of the combined regimen. A total of 102 patients were planned for enrollment in this study. This trial was expected to start in March 2021, and the end of recruitment will be approximately on March 2024, and the end of follow-up will be approximately on October 2023. The control group would take apatinib monotherapy regimen, with 500mg oral apatinib every day, and the experimental group would take apatinib plus camrelizumab regimen, with 250 mg oral apatinib every day continuously and 200mg intravenous camrelizumab every 14 days. Patients would be assessed every 8 weeks and those patients with disease control would be received the treatment until progressive disease (PD) or intolerable toxicity. The maximum treatment duration of camrelizumab was 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18;
2. Locally advanced or recurrent/metastatic gastric or gastroesophageal junction adenocarcinoma confirmed by histopathological examination;
3. Standard treatment failure of no less than two lines of systematic treatment (treatment failure is defined as intolerance of toxic and side effects, disease progression during treatment or recurrence after treatment);
4. With one or more measurable lesions, the longest diameter measured by spiral CT scan should be at least 10 mm, and the longest diameter measured by conventional CT scan should be at least 20 mm (RECIST standard, version 1.1);
5. ECOG score was 0-2;
6. Life expectancy ≥12 weeks;
7. The patient has recovered from damage caused by other anti-tumor therapy, received cytotoxic drugs, radiotherapy or surgery for ≥4 weeks, and the wound has completely healed;
8. Bone marrow capacity and liver and kidney function were sufficiently reserved 7 days before screening: absolute neutrophil (ANC) count ≥1.5x109 /L; Hemoglobin ≥ 8.0g/ dL; Platelet count ≥80 x109 /L; Total bilirubin < 1.5 times upper normal limit (ULN); ALT and AST< 2.5x ULN (with liver metastasis <5x ULN); Serum creatinine ≤1 x ULN, the clearance rate of endogenous creatinine >50ml/min;
9. Women of childbearing age should take effective contraceptive measures;
10. Subjects voluntarily joined the study and signed informed consent with good compliance and follow-up.

Exclusion Criteria:

1. A history of other malignant tumors within 5 years, except cured cervical carcinoma in situ or basal cell carcinoma of the skin;
2. Patients with hypertension that could not be controlled by antihypertensive medication (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg), coronary heart disease of grade I or above, arrhythmia of grade I or above (including prolonged QTc interval > 450ms in males and > 470 ms in females) and cardiac dysfunction of grade I or above;
3. Symptomatic brain or meningeal metastases (unless the patient was treated for >6 months, imaging results were negative within 4 weeks prior to study entry, and tumor-related clinical symptoms were stable at study entry);
4. with a history of uncontrolled epileptic seizures, central nervous system dysfunction, or mental disorders;
5. Uncontrolled pleural or abdominal effusion;
6. Undergoing kidney dialysis;
7. severe or uncontrolled infection;
8. pregnant or lactating women who are fertile but have not taken adequate contraceptive measures;
9. Multiple factors affecting oral medication (inability to swallow, chronic diarrhea and intestinal obstruction);
10. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg< 2G /L), bleeding tendency or receiving thrombolytic or anticoagulant treatment;
11. patients with gastrointestinal bleeding risk should not be enrolled, including the following conditions :(1) active peptic ulcer lesions and fecal occult blood (++); (2) patients with history of black stools and hematemesis within 3 months;
12. Prior exposure to any anti-PD-1 or anti-PD-L1, PD-L2, CD137, CTLA-4 antibody therapy, or any other antibody or drug that specifically targets T-cell costimulation or immune checkpoint pathways.
13. Participated in clinical trials of other drugs within four weeks
14. Urine routine examination indicated urine protein > 2+
15. Received systemic systemic therapy with anti-tumor indications of Chinese herbal medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, etc.) within 2 weeks before the first administration;
16. Use of immunosuppressive agents within 4 weeks prior to the first dose of study therapy, excluding nasal, inhaled, or other topical or physiological doses of systemic glucocorticoids (i.e., no more than 10 mg/ d of prednisone or equivalent doses of other glucocorticoids), or hormone use for the prevention of contrast agent allergy.
17. Residual liver volume is less than 50% of the total liver volume.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
PFS | Time Frame: from the time signing of ICF until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  progression free survival

SECONDARY OUTCOMES:
OS | from the time signing of ICF until the date of death from any cause, assessed up to 36 months
  overall survival
DoR | the time between the first tumor evaluation for CR or PR and the first evaluation for PD(Progressive Disease) or death from any cause, assessed up to 36 months
  duration of response
ORR | the rate of patients with CR and PR, through study completion, an average of 1 year
  objective response rate
DCR | the rate of patients with CR, PR and SD, through study completion, an average of 1 year
  disease control rate
AEs | the adverse events rate and types of all enrolled patients, through study completion, an average of 1 year
  the adverse events of all enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No